CLINICAL TRIAL: NCT05839145
Title: Home Monitoring of Adult Patients With SMA: a Pilot Multicenter Validation Study
Acronym: SMA-AtHome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut de Myologie, France (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SMA-AtHome
Record Dates: First submitted 2022-12-02; First posted 2023-05-03 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Muscular Atrophy, Spinal, Type II; Muscular Atrophy, Spinal, Type III
Keywords: Muscular Atrophy, Spinal; Home monitoring; BioImpedance
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Muscular Atrophy, Spinal | interventions — LIMS1 protein, human; Bleeding Time; Surveys and Questionnaires; Accelerometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home to onsite monitoring (Other): Patients will be monitored and evaluate in a first time at home then onsite.
  Interventions: Other: Strength force measurment; Other: Time tests; Other: Motor scales; Other: Questionnaires; Device: Accelerometry; Other: MNR; Other: Bio-impedance analysis
- Onsite to Home monitoring (Other): Patients will be monitored and evaluate in a first time onsite then at home .
  Interventions: Other: Strength force measurment; Other: Time tests; Other: Motor scales; Other: Questionnaires; Device: Accelerometry; Other: MNR; Other: Bio-impedance analysis

INTERVENTIONS:
Other: Strength force measurment — The grip and pinch strength of the patient will be evaluate using dedicated devices (MyoGrip and MyoPinch)
  Other Names: MyoGrip/Pinch
Other: Time tests — Lower and upper limb capacities of the patients will be measured during timed tests
  Other Names: 10mWT, 30STS, 6MWT, 9HPT
Other: Motor scales — Patient's motor functional abilities will be evaluated using specific motor scales (MFM32, RULM)
Other: Questionnaires — Patients and caregivers quality of life will be measured with different questionnaires (SMA-FRS, QOL-gNMD, SMAIS, PREM)
Device: Accelerometry — Patients physical activity will be measured at home using accelerometer sensors
Other: MNR — Sub-group of patients will perform an NMR imaging to evaluate the intramuscular fatty infiltration in thighs and muscle volume in thighs
Other: Bio-impedance analysis — The patients' muscular and fatty volume will be evaluated using BIA technic (compared to MNR)

SUMMARY:
There is no complete cure for SMA yet. However, the discovery of the genetic cause of SMA has led to the development of several treatment options that affect the genes involved in SMA - a gene replacement therapy called Zolgensma, and two drugs, called Nusinersen (Spinraza) and Risdiplam (Evyrsdi). In this context, the evaluation of efficacy and the long term follow-up of patients treated with these innovative treatments in clinical routine is one of the critical points. These evaluations are carried out in a medical context (clinical sites or research unit) using validated measurement tools and outcome measures. Carrying out these evaluations in a controlled environment can be considered from certain aspects as an advantage (reproducibility of measures, neutral environment, etc.), but also raises a certain number of questions regarding the impact on patients, the financial cost, or the relevance of the data obtained in an unnatural environment (stress, fatigue, patient motivation…). Also the regulatory authorities ask for longitudinal data for deciding to reimburse these expensive treatments. As such, the hospital cannot digest all these evaluations due to a lack of resources.

DETAILED DESCRIPTION:
In the last few years, a number of therapeutic approaches have targeted a possible increase of the production of SMN protein in target motor neurons by genetic replacement of the defective SMN1 gene or by modifying pre-mRNA splicing in SMN2 to promote exon 7 inclusion by using an antisense oligonucleotide or small molecule drugs. Several clinical studies have focused on the evaluation of patients with SMA, whether they are ambulatory or not, adults, children or infants, treated or untreated.

Depending on the SMA type, age or ambulatory status of the patients, different assessments (motor function scales or questionnaires) have provided consistent results to measure the evolution of the patients, such as HFMSE, MFM, RULM, 6MWT, MRC scale, Chop Intend or HINE.

As these evaluations are generally carried out in a controlled environment, they are likely to present an environmental bias. Even if studies are designed to anticipate and avoid most of these issues, different factors can influence patient test results (fatigue, motivation, stress, day to day variability…). From an economical point of view, the evaluation of patients in a controlled environment also has a significant cost, which heavily impact the global cost of clinical research or standard care (transport, patients' accommodation and care…). This factor is even more important as a significant proportion of the SMA population is non-ambulatory.

New treatments are indicated to treat SMA with a major impact on pre-existing disease standards of care and patients care pathway. In particular, there is no consensus on appropriate measures to monitor disease progression and treatment effect in a real-world setting. Such measures are critically needed to discuss treatment indication (treatment initiation criteria and stopping rules, therapeutic goals) and treatment monitoring. While patient reported outcome measures (PROMs) become more represented, objective functional measures are still required to assess SMA. In spite of the development of digital measures, no validated patient self-reported functional measures can be used as a surrogate. Thus, the objective disease assessment is currently based on validated outcome measures for SMA, similar to those used in clinical studies. As compared to clinical trials, the feasibility to administer these measures to SMA patients is challenging. Major limiting factors are: (1) the high disease-prevalence, (2) time-consuming measures, (3) the need for trained expert evaluators, and (4) limited access to hospital-based resources. In addition, the burden of affected individuals and caregivers has not been evaluated as well as patient treatment monitoring expectations. A refined approach using modern tools and fitting with patient real life environment is needed.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Confirmed SMA type 2 or 3 diagnostic
* Written informed consent
* Able to comply with all protocol requirements
* Affiliate or beneficiary of a social security scheme

Non-Inclusion Criteria:

* Inability to carry out assessments at home
* Claustrophobia (only for patients from Paris and Lille sites)
* Guardianship/trusteeship
* Pregnant or nursing women

Exclusion criteria:

* Inability to comply with protocol requirements
* Any medical and social conditions that could interfere with the study under the appreciation of the medical coordinator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
To compare the results of physical evaluations between home and hospital | Through study completion, an average of 3 weeks
  Evaluation of the correlations between results obtained during the physical evaluations at home compared to those obtained at hospital

SECONDARY OUTCOMES:
To determine the barriers for evaluation at home | Through study completion, an average of 3 weeks
  Inventory of items and assessments not carried out at home due to the environment
Correlation of home and hospital muscle volume measurement methods | Through study completion, an average of 3 weeks
  Comparison of muscle volumes measured by bio-impedancemetry with those obtained by MRI.
Correlation of home and hospital MyoGrip measurement | Through study completion, an average of 3 weeks
  Comparison of MyoGrip measurements obtained at home and at the hospital.
Correlation of home and hospital MyoPinch measurement | Through study completion, an average of 3 weeks
  Comparison of MyoPinch measurements obtained at home and at the hospital.
Correlation of home and hospital MFM results | Through study completion, an average of 3 weeks
  Comparison of MFM evaluation results obtained at home and at the hospital.
Correlation of home and hospital RULM results | Through study completion, an average of 3 weeks
  Comparison of RULM evaluation results obtained at home and at the hospital.
Correlation of home and hospital 30STS tests results | Through study completion, an average of 3 weeks
  Comparison of 30STS measurements obtained at home and at the hospital.
Correlation of home and hospital 9HPT results | Through study completion, an average of 3 weeks
  Comparison of 9HPT measurements obtained at home and at the hospital.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU d'Angers, Angers
  - CHU de Lille, Lille
  - CHU de Nantes, Nantes
  - Institute of Myology, Paris
  - CHU de Reims, Reims
  - CHRU de Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided